CLINICAL TRIAL: NCT07126496
Title: Precision Clinical Trial Recruitment to Promote Cancer Health Equity Across Florida (Aims 2 & 3)
Brief Title: A Virtual Community Health Educator for Increasing Clinical Trial Referrals Among Cancer Patients and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-013379; NCI-2025-05254 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-013379 (Other: Mayo Clinic Institutional Review Board); U01CA274970 (NIH)
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (ALEX Research Portal, vCHE) (Experimental): Participants receive information about available cancer clinical trials via the ALEX Research Portal and vCHE over 20-30 minutes on study.
  Interventions: Other: Questionnaire Administration; Other: Virtual Technology Intervention
- Arm II (online text) (Active Comparator): Participants receive information about available cancer clinical trials via online text on study.
  Interventions: Other: Internet-Based Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Receive information via online text
  Arms: Arm II (online text)
Other: Questionnaire Administration — Ancillary studies
Other: Virtual Technology Intervention — Receive information via ALEX Research Portal and vCHE
  Other Names: Virtual Reality Intervention; Virtual Technology
  Arms: Arm I (ALEX Research Portal, vCHE)

SUMMARY:
This clinical trial studies how well a virtual community health educator (vCHE) works in increasing clinical trial referrals for patients with cancer and their caregivers. Low enrollment of underrepresented and underserved populations in cancer clinical trials has led to disparities in intervention development and implementation. One approach to recruiting diverse populations to cancer clinical trials is community health educators. However, community health educator interventions are costly and difficult to implement. vCHEs are photo-realistic virtual agents that provide personalized guidance and support to users. They are designed to mimic real-life community health workers, offering culturally and linguistically tailored information to users. They can communicate in English or Spanish and are available in diverse genders and racial/ethnic backgrounds. vCHEs may be able to increase the enrollment of diverse participants into cancer clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Individuals Diagnosed with Cancer

  * 18 years or older
  * Must have received a cancer diagnosis at any point in your life
  * Able to understand English or Spanish
* Care Partners

  * Must be a care partner (also known as caregiver, carer, supporter, helper, aide, assistant, companion, attendant, advocate, or family caregiver) of an adult who has received a cancer diagnosis
  * Must be actively involved in the decision-making process OR care of a person diagnosed with cancer
  * Must be 18 years or older

Exclusion Criteria:

* Self-reported: people who are currently or have been in a cancer clinical trial within the last 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of referrals to cancer clinical trials (CCTs) | Up to 3 months
  Assessed by the number of referrals (patient self-referral or care partner referral) to an open cancer clinical trial (CCT).
Number of patient referrals sent by a healthcare provider by using the ALEX portal | Up to 3 months
  Assessed by the number of referral sent by providers on a patient's behalf to a study coordinator for screening.

CONTACTS AND LOCATIONS:
Overall Officials: Janice L. Krieger, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials